CLINICAL TRIAL: NCT03789357
Title: Prevalence of Primary Aldosteronism in Patients With Stroke
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PA_CVA
Record Dates: First submitted 2018-12-19; First posted 2018-12-28 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Primary Aldosteronism; Stroke
Keywords: Hypertension; Arrhythmia; Adrenal vein sampling; Mineralocorticoid-receptor Antagonists
MeSH Terms: conditions — Hyperaldosteronism; Stroke; Hypertension; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: All patients admitted to the Acute Stroke Unit
  Interventions: Diagnostic Test: Aldosterone renin ratio

INTERVENTIONS:
Diagnostic Test: Aldosterone renin ratio — Aldosterone Renin Ratio to screen for Primary Aldosteronism

SUMMARY:
Strokes leads to significant morbidity and mortality, and hypertension is the most important risk factor for strokes. It is estimated that up to 10% of patients with hypertension have the underlying, treatable condition of primary aldosteronism. Hence, we hypothesize that the prevalence of primary aldosteronism is high in patients with strokes, a complication of long-standing hypertension.

Patients admitted with an acute stroke to the Acute Stroke Unit, Changi General Hospital, will be screened for Primary Aldosteronism three months post-stroke, and confirmatory tests will be done with saline-infusion test.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-80 years
2. Admitted with acute cerebrovascular accident (CVA) or transient ischemic attack (TIA) to the ASU, CGH
3. Patients with both ischemic and hemorrhagic strokes

Exclusion Criteria:

a. Pregnant patients

Ages: 21 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective study to evaluate the prevalence of primary aldosteronism in patients with an acute stroke. 300 patients admitted with CVA/TIA will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with stroke with confirmed primary aldosteronism in patients admitted to the acute stroke unit for stroke | 6 months
  Percentage of patients with confirmed Primary Aldosteronism using confirmatory test

SECONDARY OUTCOMES:
Accuracy of Screening test in early period post-stroke | 3 months
  To determine if the screening blood test for primary aldosteronism performed within 1 week post-stroke is equally accurate compared to being performed 2-4 months post-stroke.
Percentage of unilateral primary aldosteronism in patients admitted with acute stroke | 6 months
  Percentage of unilateral PA amongst patients with stroke
Percentage of patients with positive screening test in patients admitted with acute stroke | 3 months
Blood pressure change after treatment for primary aldosteronism | 12 months
Cardiac Complications | 6 months
  Cardiac complications in patients with primary aldosteronism, compared to those without primary aldosteronism, as assessed by transthoracic echocardiography features of left ventricular hypertrophy / mass, and diastolic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Troy Puar, MRCP UK, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen V, Tu TM, Mamauag MJB, Lai J, Saffari SE, Aw TC, Ong L, Foo RSY, Chai SC, Fones S, Zhang M, Puar TH. Primary Aldosteronism More Prevalent in Patients With Cardioembolic Stroke and Atrial Fibrillation. Front Endocrinol (Lausanne). 2022 Apr 19;13:869980. doi: 10.3389/fendo.2022.869980. eCollection 2022. PMID 35518929